CLINICAL TRIAL: NCT00006104
Title: A Multi-Institutional Phase II Pilot Trial With Weekly Docetaxel and Herceptin as First or Second Line Therapy for HER2/Neu Overexpressing Metastatic Breast Cancer
Brief Title: Trastuzumab Plus Docetaxel in Treating Women With Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Purpose: Treatment
Other Study IDs: VICC BRE 9823; P30CA068485 (NIH); VU-VCC-BRE-9823; NCI-G00-1830
Record Dates: First submitted 2000-08-03; First posted 2003-12-24 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: trastuzumab
Drug: docetaxel

SUMMARY:
RATIONALE: Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of trastuzumab plus docetaxel in treating women who have recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate of women with HER2-neu overexpressing recurrent or metastatic breast cancer treated with trastuzumab (Herceptin) in combination with docetaxel. II. Determine the toxicity of this treatment regimen in these patients. III. Determine the duration of response to this treatment regimen in these patients. IV. Determine the time to progression in these patients after receiving this treatment regimen. V. Compare HER2-neu overexpression as determined by fluorescent in situ hybridization (FISH) versus immunohistochemistry, and correlate these findings with response to this treatment regimen in these patients. VI. Correlate HER2-neu activation by immunohistochemistry and the extracellular domain of HER2-neu by ELISA with response to this treatment regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive docetaxel IV over 30 minutes weekly for 6 weeks plus trastuzumab (Herceptin) IV over 30-90 minutes weekly for 8 weeks. Treatment continues every 8 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed monthly for 3 months, every 3 months for 9 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 18-34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or metastatic breast cancer HER2-neu overexpressing tumor (2+ or 3+) Measurable or evaluable disease If bone disease only, must have lytic lesions No carcinomatous meningitis or untreated or uncontrolled brain parenchymal disease Prior brain parenchymal disease allowed if controlled by appropriate therapy given at least 8 weeks prior to study, and patient is asymptomatic from CNS disease Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal Alkaline phosphatase no greater than 2.5 times upper limit of normal (ULN) SGOT and SGPT no greater than 1.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No congestive heart failure Ejection fraction greater than 45% by MUGA No myocardial infarction within the past 6 months No ischemic heart disease requiring medication No uncontrolled hypertension Other: No peripheral neuropathy grade 2 or more No other prior malignancy within the past 5 years except curatively treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or contralateral breast cancer No active unresolved infection No history of hypersensitivity reaction to products containing Polysorbate 80 No poorly controlled diabetes mellitus Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic response modifiers Chemotherapy: Prior adjuvant chemotherapy allowed No more than 1 prior chemotherapy regimen for metastatic disease No prior taxane (docetaxel or paclitaxel) Prior doxorubicin allowed if total dose less than 250 mg/m2 No other concurrent chemotherapy Endocrine therapy: Prior hormonal therapy allowed No concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy No prior cumulative radiotherapy to more than 25% of bone marrow No concurrent radiotherapy Surgery: Not specified Other: At least 7 days since prior antibiotics No other concurrent investigational drugs No other concurrent antineoplastic therapy No concurrent parenteral antibiotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1998-09; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (15):
- United States (15):
  - Providence Hospital, Mobile, Alabama
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Owensboro Medical Health System, Owensboro, Kentucky
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Erlanger Health Systems, Chattanooga, Tennessee
  - Memorial Health Care System, Chattanooga, Tennessee
  - Williamson Medical Center, Franklin, Tennessee
  - Jackson-Madison County Hospital, Jackson, Tennessee
  - Methodist/Thompson Oncology Research, Knoxville, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Boston Baskin Cancer Group, Memphis, Tennessee
  - St. Thomas Health Services, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Methodist Medical Center of Oak Ridge, Oak Ridge, Tennessee